CLINICAL TRIAL: NCT02163811
Title: Self-management to Improve Function Following Amputation
Acronym: VETPALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Spectrum Research, Inc. (Industry); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: D1143-R
Record Dates: First submitted 2014-06-05; First posted 2014-06-16 (Estimated); Results first posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Amputation, Limb Loss
Keywords: Self-management; Functional status; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VETPALS (Experimental): VETPALS is a five session course utilizing adult learning methods to teach self-management for people with life changes after amputation. The five sessions are held weekly, and are facilitated by a VA Puget Sound clinician in conjunction with a peer facilitator (Veteran with limb loss).
  Interventions: Behavioral: VETPALS
- Individual Education Support Program (Active Comparator): VETPALS facilitator provide post-amputation education materials from the Amputee Coalition, including First Step - A Guide for Adapting to Limb Loss and Side Step - A Guide to Preventing and Managing Diabetes and Its Complications. Veterans receive all usual care.
  Interventions: Behavioral: Individual Education Support Program

INTERVENTIONS:
Behavioral: VETPALS — VETPALS is an adaption of an empirically supported self-management program, PALS (Promoting Amputee Life Skills). The PALS program demonstrated improved physical and psychosocial functioning when delivered in community-based support groups for amputees, but this program has not been adapted for the needs of Veterans and implemented in the VA healthcare system.
  VETPALS is a five session course for people with life changes after amputation. The five sessions are held weekly, and are facilitated by a VA clinician in conjunction with a peer facilitator (Veteran with limb loss). Veterans receive all usual care.
  Arms: VETPALS
Behavioral: Individual Education Support Program — VETPALS facilitator provide post-amputation education materials from the Amputee Coalition, including First Step - A Guide for Adapting to Limb Loss and Side Step - A Guide to Preventing and Managing Diabetes and Its Complications. Veterans receive all usual care.
  Arms: Individual Education Support Program

SUMMARY:
Lower extremity amputations are a significant cause of morbidity, mortality, loss of function and reduced quality of life. Self-management (defined as the process by which an individual adopts an active role in managing the symptoms, treatment, consequences, and lifestyle changes inherent in living with a chronic condition) is an important mechanism for improving health and reducing disability. This study will evaluate a 5-week group-based self-management intervention for Veterans with lower extremity limb loss (VETPALS) and determine its impact upon physical and psychosocial functioning, patient activation, self-efficacy, problem solving, quality of life and positive affect. This study represents one of the only prospective randomized controlled trials of a behavioral intervention for individuals with limb loss. It is expected that results will be used to inform the integration of self-management interventions into the VA Amputation System of Care. The specific primary hypotheses are:

1. Individuals randomized to VETPALS will display greater improvements from baseline in physical functioning as measured by the MFA-SF than Veterans in the individual education support condition post-intervention and at a 6 month follow-up.
2. Individuals randomized to VETPALS will display greater improvements from baseline in psychosocial functioning as measured by the PHQ-9 than Veterans in the individual education support condition post-intervention and at a 6 month follow-up.

DETAILED DESCRIPTION:
Self-management interventions have been successful in improving outcomes across a broad variety of chronic illnesses including arthritis, asthma, diabetes, and hypertension. Initial evidence of the effectiveness of self-management following limb loss is promising, but limited. Only one published trial to date has examined self-management for amputees. The Promoting Amputee Life Skills (PALS) project, conducted by members of the current study team, designed and implemented an 8-week group-based intervention to improve self-management following limb loss. The current proposal builds upon previous research that has demonstrated the efficacy of the PALS self-management intervention, but addresses important next questions:

1. Is the PALS self-management intervention appropriate for Veterans, specifically considering the very high prevalence of diabetes and vascular disease?
2. Can it be housed and delivered within a health care system as opposed to existing community support groups?
3. Will the intervention be more effective for individuals who are new amputees?
4. Will a shorter format that also incorporates an option for video teleconferencing retain the efficacy of the original PALS intervention?

This study is a two-arm randomized controlled trial (RCT) to determine the efficacy of VETPALS. Study staff will screen and enroll Veterans with recent lower extremity limb loss within the last 6 months. Each participant will complete a baseline interview and then is sequentially placed into a cohort of 6-10 participants; each cohort will be randomized to the VETPALS group based self-management program (intervention) or an individual education support program (control). Once participants complete the randomized arm and follow-up assessments, they are free to participate in the other group. This ensures participants are offered both programs and are not deprived of a potentially valuable healthcare service.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 or older
* Has had transmetatarsal amputation (through the foot including Chopart and Lisfranc amputation), transtibial amputation (below the knee), transfemoral amputation (above the knee), knee disarticulation (at knee), or hip disarticulation (at hip) due to dysvascular disease/diabetes. These can all include a revision of an amputation.
* Participant has a contact address and phone number so that s/he can be reached during the course of the study.*
* Enrolled within 6 months of amputation.
* Speak and comprehend English.

  * The investigators will ask a participant who does not meet eligibility criteria because of inclusion criteria item 3 if s/he will have one in the near future, and if yes, permission to contact them again at that time. This allows the participant to be included, if interested and eligible, at a later date.

Exclusion Criteria:

* Inadequate cognitive or language function to consent or participate defined by greater than or equal to 6 errors on the SPMSQ or diagnosis of dementia or Alzheimer's disease.
* Active substance use disorder identified by chart review and initial screening. Note: No personnel involved in the study may identify, directly or indirectly, any individual patient or participant in any report of such research or otherwise disclose patient or participant identities in any manner.
* Major uncontrolled psychiatric illness (bipolar disorder, psychosis, severe suicidality) identified by chart review and confirmed as necessary by discussion with current providers.
* Spinal Cord Injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron P Turner, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA; Gail Latlief, DO, Principal Investigator — James A. Haley Veterans' Hospital, Tampa, FL; Samuel L. Phillips, PhD, Principal Investigator — James A. Haley Veterans' Hospital, Tampa, FL
Locations (5):
- United States (5):
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turner AP, Wegener ST, Williams RM, Ehde DM, Norvell DC, Yanez ND, Czerniecki JM, Study Group V. Self-Management to Improve Function After Amputation: A Randomized Controlled Trial of the VETPALS Intervention. Arch Phys Med Rehabil. 2021 Jul;102(7):1274-1282. doi: 10.1016/j.apmr.2021.02.027. Epub 2021 Apr 1. PMID 33811854
- See also: Click here for more information about this study: Self-management to Improve Function Following Amputation — http://www.amputee-coalition.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 182 enrolled 147 were randomized
Pre-assignment Details: 9 Deaths, 26 withdrawal
Groups:
- Individual Education Support Program: Individual Education Support Program: VETPALS facilitator provides post-amputation education materials from the Amputee Coalition and offer for individual follow-up for explanation if requested. Veterans receive all usual care.
Period: Overall Study
Arm/Group | VETPALS | Individual Education Support Program
Started | 71 | 76
Completed | 35 | 60
Not Completed | 36 | 16

BASELINE CHARACTERISTICS:
Population: Individuals with Limb Loss Randomized to VETPALS or Education Control
Groups:
- Total: Total of all reporting groups
Arm/Group | VETPALS | Individual Education Support Program | Total
Number analyzed (Participants) | 71 | 76 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.89 (8.34) | 64.12 (8.55) | 64.49 (8.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 68 | 76 | 144
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 25 | 18 | 43
  White | 44 | 50 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 7
Marital Status (Married) [Count of Participants; unit: Participants] | 32 | 26 | 58
Education [Mean (Standard Deviation); unit: years] | 13.44 (2.2) | 13.96 (2.26) | 13.71 (2.24)
Months since amputation [Mean (Standard Deviation); unit: Months] | 10.49 (7.32) | 9.62 (5.54) | 10.04 (6.45)
Amputation Level [Count of Participants; unit: Participants]
  Transmetatarsal | 3 | 8 | 11
  Transtibial | 53 | 57 | 110
  Transfemoral | 15 | 11 | 26
Comorbidity [Mean (Standard Deviation); unit: comorbidities] | 4.90 (2.71) | 4.11 (2.36) | 4.49 (2.55)
Mental Status [Mean (Standard Deviation); unit: units on a scale] — Short Portable Mental Status Questionnaire, range 0-10, higher scores indicating better function
  units on a scale | 9.73 (.54) | 9.62 (.71) | 9.67 (.63)
Physical Functioning [Mean (Standard Deviation); unit: units on a scale] — Short Musculoskeletal Functional Assessment dysfunction index, range = 0-100 with higher scores indicating poorer function.
  units on a scale | 33.17 (16.19) | 29.14 (15.35) | 31.09 (15.84)
Psychosocial Functioning [Mean (Standard Deviation); unit: units on a scale] — Patient Health Questionnaire depression module (PHQ-9). Scores range from 0 to 27 with higher scores indicating higher levels of depression
  units on a scale | 6.08 (5.75) | 4.22 (4.37) | 5.12 (5.15)
Pain [Mean (Standard Deviation); unit: units on a scale] — Chronic Pain Grade Pain Intensity. Range = 0-100 with higher values reflecting higher levels of pain intensity
  units on a scale | 47.75 (25.48) | 41.75 (27.13) | 44.65 (26.43)
Quality of Life [Mean (Standard Deviation); unit: units on a scale] — World Health Organization Quality of Life Scale (WHOQoL-BREF): Overall quality of life. Range = 1-5 with higher scores indicating higher QoL
  units on a scale | 3.69 (.98) | 3.87 (.90) | 3.78 (.94)
Satisfaction with Health [Mean (Standard Deviation); unit: units on a scale] — World Health Organization Quality of Life Scale (WHOQoL-BREF): Satisfaction with Health. Range = 1-5 with higher scores indicating higher satisfaction with health.
  units on a scale | 3.30 (.98) | 3.64 (1.09) | 3.48 (1.05)
Social Support (MSPSS) [Mean (Standard Deviation); unit: units on a scale] — Multidimensional Scale of Perceived Social Support. Range = 1-7 with higher values indicating higher levels of social support
  units on a scale | 5.25 (1.38) | 5.39 (1.47) | 5.33 (1.42)
Self-Efficacy [Mean (Standard Deviation); unit: units on a scale] — Measure of self-efficacy. Range = 0-10 with higher levels indicating higher levels of self-efficacy
  units on a scale | 7.72 (2.12) | 8.14 (1.71) | 7.94 (1.93)
Patient Activation Measure [Mean (Standard Deviation); unit: units on a scale] — Measure of patient engagement and activation in health and self care. Range = 1-5 with higher values representing greater patient activation.
  units on a scale | 3.01 (.73) | 3.21 (.75) | 3.12 (.75)
Social Problem Solving Inventory [Mean (Standard Deviation); unit: units on a scale] — Measure of problem solving. Range 0-100 with higher scores representing better problem solving
  units on a scale | 72.56 (15.83) | 77.27 (14.20) | 74.99 (15.14)
Positive and Negative Affect Scale (PANAS) Positive Affect Score [Mean (Standard Deviation); unit: units on a scale] — Positive Affect Subscale. Range = 10 to 50. Higher values represent greater positive affect
  units on a scale | 31.83 (9.15) | 33.57 (9.84) | 32.73 (9.52)

OUTCOME MEASURES:

1. Primary Outcome: Short Musculoskeletal Function Assessment (SMFA)
Description: Physical functioning will be measured using the Short Musculoskeletal Function Assessment (SMFA) Dysfunction Index. Range = 0 - 100 with higher values reflecting poorer physical function
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VETPALS | Individual Education Support Program
Number analyzed (Participants) | 35 | 60
score on a scale | 32.34 (17.85) | 30.19 (19.42)

2. Primary Outcome: Patient Health Questionnaire (PHQ-9)
Description: Psychosocial functioning will be evaluated by examining depression using the Patient Health Questionnaire Depression Module (PHQ-9). Range = 0-27 with higher scores indicating greater levels of depression
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VETPALS | Individual Education Support Program
Number analyzed (Participants) | 35 | 60
score on a scale | 5.14 (4.83) | 5.87 (6.23)

3. Secondary Outcome: World Health Organization Quality of Life Scale (WHOQOL-BREF) Overall Quality of Life
Description: Overall Quality of Life Scale. Range = 1-5 with higher values reflecting better quality of life.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VETPALS | Individual Education Support Program
Number analyzed (Participants) | 35 | 60
score on a scale | 3.86 (.88) | 3.77 (1.13)

4. Secondary Outcome: World Health Organization Quality of Life Scale (WHOQOL-BREF) Satisfaction With Health
Description: Satisfaction with Health Scale. Range = 1 to 5. Higher values represented better satisfaction with health
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VETPALS | Individual Education Support Program
Number analyzed (Participants) | 35 | 60
score on a scale | 3.69 (.96) | 3.32 (1.38)

5. Other Pre Specified Outcome: Self-Efficacy
Description: Self-Efficacy for self-management of limb loss. Range = 0 to 10. Higher values reflect greater self-efficacy
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VETPALS | Individual Education Support Program
Number analyzed (Participants) | 35 | 60
score on a scale | 7.96 (1.78) | 7.89 (2.15)

6. Other Pre Specified Outcome: Patient Activation Measure
Description: Participant Active Engagement in Self-Care. Range = 1 to 5. Higher values reflect greater active engagement.
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VETPALS | Individual Education Support Program
Number analyzed (Participants) | 35 | 60
score on a scale | 3.17 (.92) | 3.08 (.99)

7. Other Pre Specified Outcome: Social Problem Solving Inventory
Description: Active Problem Solving. Range = 0 to 100. Higher values represent greater problem solving
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VETPALS | Individual Education Support Program
Number analyzed (Participants) | 35 | 60
score on a scale | 72.06 (15.35) | 76.29 (16.21)

8. Other Pre Specified Outcome: Positive and Negative Affect Scale (PANAS) Positive Affect Score
Description: Positive Affect Subscale. Range = 10 to 50. Higher values represent greater positive affect.
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VETPALS | Individual Education Support Program
Number analyzed (Participants) | 35 | 60
score on a scale | 32.69 (9.94) | 31.38 (10.04)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | VETPALS | Individual Education Support Program
All-Cause Mortality (participants affected / at risk) | 6/71 | 2/76
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/76
Other Adverse Events (participants affected / at risk) | 0/71 | 0/76

LIMITATIONS AND CAVEATS:
Results based on a sample of individuals with dysvascular disease/diabetes and may not generalize to all amputees.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT02163811/Prot_SAP_000.pdf